CLINICAL TRIAL: NCT01534377
Title: Prevention of Depression in Maltreated and Nonmaltreated Adolescents
Brief Title: Interpersonal Psychotherapy for Adolescent Girls
Acronym: IPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Sheree Toth, Director Mt. Hope Family Center, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 035457; 1R01MH091070-01A1 (NIH)
Record Dates: First submitted 2012-02-02; First posted 2012-02-16 (Estimated); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Depression
Keywords: Depression; Adolescents
MeSH Terms: conditions — Depression | interventions — Interpersonal Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Interpersonal Psychotherapy (Experimental): Adolescents will receive Interpersonal Psychotherapy for the treatment and prevention of depression.
  Interventions: Behavioral: Interpersonal Psychotherapy for Adolescents
- Enhanced Care (Experimental): Adolescents will receive the Enhanced care model or care that they would typically receive in community setting to treat and prevent depression.
  Interventions: Behavioral: Enhanced Care

INTERVENTIONS:
Behavioral: Interpersonal Psychotherapy for Adolescents — Adolescents will receive IPT-A a manualized intervention for depression and prevention of depression that emphasizes current interpersonal relationships, focusing on their immediate social context.
  Other Names: IPT-A
  Arms: Interpersonal Psychotherapy
Behavioral: Enhanced Care — Adolescents will receive enhanced care which is consistent with care typically provided in community settings to treat and prevent depression.
  Other Names: EC
  Arms: Enhanced Care

SUMMARY:
This study will evaluate the efficacy of Interpersonal Psychotherapy for Adolescents (IPT-A) for the treatment of depression and prevention of depression in maltreated and nonmaltreated girls between the ages of 13-15 years old.

DETAILED DESCRIPTION:
Child maltreatment poses a serious public health problem and heightens the risk of psychopathology across the life course. Adolescence also represents a peak time for the emergence of depressive disorders particularly in girls. Effective interventions to prevent and treat depression in low income adolescent girls with or without histories of maltreatment are needed.

Three groups will be recruited: Maltreated Depressive Symptoms (MDS), Nonmaltreated Depressive Symptoms (NDS), and a Nonmaltreated Nonsymptomatic Comparison (NNC), comparable in SES, race/ethnicity, and household composition. The MDS and NDS groups will be randomized into IPT-A or Enhanced Care (EC). Adolescent girls in these groups will receive 13 sessions of therapy. Girls in the NNC group will only complete research visits.

Research assessments will be conducted at T1 (baseline/prior to intervention), T2 (6-weeks mid-intervention), T3 (end of intervention), T4 (1-year post) and T5 (18 months post). Girls and their mothers will participate in these research sessions. A multi-level-of-analysis approach, integrating genotyping, hormone assays, cognitive testing, adolescent- and maternal-report, mother-teen observation, and DHS and school records will be utilized to assess the effectiveness of the interventions.

ELIGIBILITY:
Inclusion Criteria:

* girls
* ages 13-15 years old
* low SES status
* live in Rochester or surrounding counties
* girls in the maltreated depressive symptom group will have CPS-documented child maltreatment
* girls in the nonmaltreated depressive symptom group will not have CPS- documented child maltreatment
* girls in the nonmaltreated nonsymptomatic comparison group will have no current or past mental illness and no documented child maltreatment

Exclusion Criteria:

* taking antidepressants or prescription medications for anxiety
* already receiving mental health treatment
* actively suicidal
* diagnosed with a severe mental disorder
* abusing drugs or alcohol
* evidence of compromised cognitive ability
* evidence of a pervasive developmental disorder
* evidence of a major physical or neurological disorder
* non-English speaking

Ages: 13 Years to 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 328 (Actual)
Dates: Start 2011-07 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Change in adolescent depressive symptoms from baseline to post-intervention | Baseline and 12 weeks, follow up at 1 year & again at 18 months post intervention
  To evaluate the efficacy of Interpersonal Psychotherapy for Adolescents (IPT-A) for decreasing depressive symptoms and preventing depression in low-income ethnically and culturally diverse adolescent girls with and without histories of child maltreatment

CONTACTS AND LOCATIONS:
Overall Officials: Sheree Toth, PhD, Principal Investigator — University of Rochester; Dante Cicchetti, Ph.D., Principal Investigator — University of Minnesota
Locations (1):
- Mt. Hope Family Center, Rochester, New York, United States